CLINICAL TRIAL: NCT07071584
Title: Evaluation of a Multi-electrode Prosthesis Control System for Real-World Tasks Performance
Brief Title: Evaluation of a Multi-electrode Prosthesis Control System for Real-world Tasks Performance in Individuals With Upper Limb Transradial Amputation
Acronym: EMPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phantom Neuro Inc. (Industry)
Collaborators: Atlas Ambulatory Surgery Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PN02
Record Dates: First submitted 2025-06-19; First posted 2025-07-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Upper Limb Amputation Below Elbow
Keywords: Myoelectric control; Transradial amputee; Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants instrumented with cutaneous version of Phantom X system using a universal socket (Experimental): With Phantom X system instrumented, participants will perform the following two assessments: ACMC and tBBT. They will also complete user satisfaction and NASA-TLX questionaries.
  Interventions: Device: Cutaneous Prosthesis Control System

INTERVENTIONS:
Device: Cutaneous Prosthesis Control System — Prosthesis control system using a multi-electrode cutaneous sensor array

SUMMARY:
This study tests how well the Phantom X prosthesis control system works. The system helps control a prosthetic hand using muscle signals from the arm. You'll wear a non-invasive version for one day in the clinic. You'll practice hand movements and then do two simple tasks with both your usual prosthesis and the Phantom X system. At the end, you'll fill out short surveys about your experience.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the functional performance of the Phantom X prosthesis control system using a non-invasive version of its 32-electrode sensor array. All other components, including the Fusion Port, will be in their final clinical form factor, consistent with those used in future implantable configurations. The study will take place during a single, in-clinic session. Informed consent will be obtained either remotely prior to the visit or at the start of the session. Participants will undergo an initial EMG screening to determine signal suitability. Those with insufficient signal quality will be excluded. Eligible participants will be fitted with a universal socket, prosthesis, and the Phantom X system. Accelerometers will be placed on both limbs for movement tracking. Participants will practice a predefined set of gestures, followed by system calibration. Two validated functional assessments, Assessment of Capacity for Myoelectric Control (ACMC) and Targeted Box and Blocks Test (tBBT), will be conducted under two conditions: with the participant's baseline setup (if applicable) and with Phantom X. The testing order will be randomized. Participants will complete a user satisfaction questionnaire and NASA Task Load Index instrument to measure intuitiveness of Phantom X system before exiting the study.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 21 years in age and older
2. Individuals with unilateral or bilateral amputation at transradial level
3. Patient is willing to comply with study protocol and make required study visits
4. Willingness and ability to sign Informed Consent

Exclusion Criteria:

1. Cognitively impaired to follow study instructions
2. Allergies to skin adhesive materials necessary for cutaneous electrode placement
3. Excessive hair growth on arms and inability to shave off the hair for electrode placement
4. Pregnant woman
5. Residual limbs of insufficient diameter or length to accommodate the wearing of two cutaneous sensor arrays
6. Injuries, bruises, or open wounds on the arm that needs to be instrumented for the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Phantom X Prosthesis Control System in performing activities of daily living (ADL) | Through study completion, average of 1 day
  Feasibility of prosthesis control will be assessed using Assessment of Capacity of Myoelectric Control (ACMC) and while participants perform predefined ADL tasks. ACMC score ranges from 0-100, higher score suggesting better prosthesis myoelectric control.
Feasibility of Phantom X Prosthesis Control System in performing repeated task requiring hand dexterity | Through study completion, average of 1 day
  Feasibility of Phantom X system in performing repeated task requiring prosthetic hand's dexterity will be assessed using Targeted Box and Blocks Test (tBBT) in which participants will transfer numbered blocks from one compartment to corresponding spots in a second adjacent compartment. tBBT is scored by measuring time taken to complete block transfer from one compartment to another. Lower completion time suggests better performance.

SECONDARY OUTCOMES:
Satisfaction of prosthesis control with Phantom X system | Through study completion, average of 1 day
  Participant satisfaction in using the Phantom X control system will be collected using a questionnaire
Intuitiveness of prosthesis control using Phantom X system | Through study completion, average of 1 day
  Intuitiveness of prosthesis control with Phantom X control system will be evaluated using NASA-Task Load Index instrument (NASA-TLX)

CONTACTS AND LOCATIONS:
Overall Officials: Elad Levy, MD, Principal Investigator — Atlas Ambulatory Surgery Center, Buffalo, NY
Locations (2):
- United States (2):
  - Atlas Ambulatory Surgery Center, Buffalo, New York
  - Phantom Neuro Inc. Operational Headquarters, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided